CLINICAL TRIAL: NCT01483040
Title: a Prospective Clinical Study to Establish the Usability of the PeerScope B System™ When Used During Standard Colonoscopy Procedure
Brief Title: PeerScope B System™ Clinical Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PeerMedical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CD-1130
Record Dates: First submitted 2011-11-22; First posted 2011-12-01 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Colon Cancer; Colon Diseases; Colon Polyps; Colon Adenomas
Keywords: wide angle view colonoscopy; PeerScope B System™
MeSH Terms: conditions — Colonic Neoplasms; Colonic Diseases; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: colonoscopy system (PeerScope B System™) — Cancer of the colon and rectum is second only to lung cancer as the leading cause of cancer-related deaths in the United States.Each year, about 1.23 million new cases of bowel cancer are diagnosed worldwide, 333,000 in Europe alone. Colorectal cancer almost always starts in a benign growth called a polyp. Polyps originate in the inner lining of the colon, where they may be visible in a screening test known as colonoscopy. Recent research has shown that appropriate screening and treatment can alleviate much of the suffering associated with colorectal cancer and reduce the number of deaths caused by this malignancy

SUMMARY:
The PeerScope B System™ by PeerMedical Ltd. is intended to provide visualization (via a video monitor) and therapeutic access to the lower intestinal tract. The lower intestinal tract includes, but is not restricted to the organs, tissues and subsystems: large bowel and cecum. The device is introduced rectally, as with any standard colonoscope when indications consistent with the need for the procedure are observed in the adult patient population.

The purpose of this prospective clinical study is to establish the usability of the PeerScope B System™ when used during standard colonoscopy procedure.

The study population is comprised of patients indicated for colonoscopy.

The primary endpoint is reaching the cecum of the colon with PeerScope B System™.Secondary endpoints:

1. The first secondary endpoint is the incidence of complications using the PeerMedical colonoscope.
2. The second secondary endpoint is successful therapeutic interventions as biopsies, polypectomies, APC etc.
3. The third secondary endpoint is the procedure time.
4. The fourth secondary endpoint is the subjective evaluation of the additional view angle by the physician.
5. The fifth secondary endpoint is patient satisfactory.

DETAILED DESCRIPTION:
Founded in 2009, PeerMedical develops colonoscopes capable of wide view angle at the press of the button. The PeerScope B System™ is an endoscopic platform that enables the physician to get a wide angle view while maintaining all of the features commonly used during Gastrointestinal (GI) procedures with very limited learning curve and in service process. The current standard devices have viewing limitations. By adding this viewing functionality, PeerMedical will potentially empower physicians to improve polyps detection and cancers within the colon.

ELIGIBILITY:
Inclusion Criteria:

* Subject between the ages of 18 and 70
* The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

* Patients with a history of colonic resection;
* Patients with inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected chronic stricture potentially precluding complete colonoscopy;
* Patients with diverticulitis or toxic megacolon;
* Patients with a history of radiation therapy to abdomen or pelvis;
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is reaching the cecum of the colon with PeerScope B S | 6 month
  a full colonoscopy procedure is characterized by reaching an anatomical mark (cecum)at the end of the insertion phase and then the physician start the withdrawal screening phase

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gralnek, Prof., Principal Investigator — Ministry of Health, Israel
Locations (1):
- Elisha Medical Center, Haifa, Israel